CLINICAL TRIAL: NCT02118922
Title: A Study to Test the Diagnostic Potential of Brillouin Microscopy for Corneal Ectasia
Status: Recruiting | Type: Observational
Sponsor: Massachusetts General Hospital (Other)
Collaborators: Harvard Medical School (HMS and HSDM) (Other)
Responsible Party: Principal Investigator, Seok Hyun Yun, Associate Professor, Massachusetts General Hospital
Other Study IDs: 2012P002178
Record Dates: First submitted 2014-04-16; First posted 2014-04-21 (Estimated); Last update posted 2025-11-06 (Actual); Status verified 2025-11

CONDITIONS: Keratoconus; Ectasia; Crosslinking; Fuchs' Endothelial Dystrophy
Keywords: LASIK
MeSH Terms: conditions — Keratoconus; Dilatation, Pathologic; Fuchs' Endothelial Dystrophy

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Cross-Sectional
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (7):
- Healthy volunteers: Volunteers with normal corneas
  Interventions: Procedure: Brillouin imaging
- Patients with keratoconus: Patients diagnosed with keratoconus
  Interventions: Procedure: Brillouin imaging
- post-LASIK no complications: Subjects who underwent LASIK refractive surgery with no complications
  Interventions: Procedure: Brillouin imaging
- post-LASIK who developed ectasia: patients who underwent LASIK refractive surgery and developed ectasia as a complications
  Interventions: Procedure: Brillouin imaging
- Volunteers to receive PRK surgery: This group includes patients who have been diagnosed with myopia and have been scheduled to undergo PRK surgery. Patients with high astigmatism > 2 diopter, prior ocular surgeries, and those patients taking any ocular medications except seasonal allergy medicine such as ketotifen or artificial tears will be excluded.
  Interventions: Procedure: Brillouin imaging
- Volunteers to receive LASIK Surgery: This group includes myopic patients who are scheduled to receive LASIK surgery. Patients with high astigmatism > 2 diopter, prior ocular surgeries, and those patients taking any ocular medications except seasonal allergy medicine such as ketotifen and artificial tears will be excluded.
  Interventions: Procedure: Brillouin imaging
- Patients with Fuch's Endothelial Corneal Dystrophy: This group includes subjects who are diagnosed with Fuch's corneal dystrophy, at early, mild and advanced stages. The inclusion also extends to subjects with, and without keratoconus. But this exclude patients with any other corneal disorders other than keratoconus, and/or history of ophthalmological surgeries that may affect endothelium cell status, e.g. cataract surgeries.
  Interventions: Procedure: Brillouin imaging

INTERVENTIONS:
Procedure: Brillouin imaging

SUMMARY:
We have developed novel Brillouin microscopy and we are testing its potential for keratoconus and ectasia diagnostics. We plan to perform axial scans of the cornea in human volunteers in order to compare biomechanical properties of Keratoconus vs. Normal corneas and compare biomechanical properties of post-LASIK ectasia vs. normal corneas.

ELIGIBILITY:
Inclusion Criteria:

Group I includes healthy subjects with normal appearing corneas, normal topography and pachymetry. Group II includes patients diagnosed as having mild, moderate or advanced keratoconus by our ophthalmology expert on the basis of topography and pachymetry. Group III includes healthy subjects who have undergone LASIK surgery in the past 12 months without complications. Inclusion criteria include normal post-operative topography and pachymetry. Group IV includes patients (age 20 - 60) who have undergone LASIK surgery at least 12 months before the study imaging and have been diagnosed with post-LASIK ectasia based on topography, pachymetry and clinical evaluation.Patients diagnosed with keratoconus. Group V- Volunteers to receive PRK surgery This group includes patients who have been diagnosed with myopia and have been scheduled to undergo PRK surgery. Patients with high astigmatism > 2 diopter, prior ocular surgeries, and those patients taking any ocular medications except seasonal allergy medicine such as ketotifen or artificial tears will be excluded. Group VI-Volunteers to receive LASIK Surgery This group includes myopic patients who are scheduled to receive LASIK surgery. Patients with high astigmatism > 2 diopter, prior ocular surgeries, and those patients taking any ocular medications except seasonal allergy medicine such as ketotifen and artificial tears will be excluded. Group VII- Patients with Fuch's Endothelial Corneal Dystrophy. This group includes subjects who are diagnosed with Fuch's corneal dystrophy, at early, mild and advanced stages. The inclusion also extends to subjects with, and without keratoconus. But this exclude patients with any other corneal disorders other than keratoconus, and/or history of ophthalmological surgeries that may affect endothelium cell status, e.g. cataract surgeries.

Overall Exclusion Criteria for all groups: Volunteers who

* Have occludable narrow angles (without a patent peripheral iridotomy)
* Monocular subjects
* Do not or cannot understand the instructions for the imaging

Ages: 20 Years to 75 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: General population
Sampling Method: Non-Probability Sample
Enrollment: 168 (Estimated)
Dates: Start 2013-06 (Actual); Primary Completion 2026-09 (Estimated); Study Completion 2026-09 (Estimated)

PRIMARY OUTCOMES:
Elastic Modulus of the Cornea | 2012-2022
  Patients will be measured one time only at their imaging session

CONTACTS AND LOCATIONS:
Overall Officials: Andy Yun, PhD, Principal Investigator — Masachusetts General Hospital
Locations (1):
- Massachusetts General Hospital, Boston, Massachusetts, United States

REFERENCES:
- [Background] Scarcelli G, Kling S, Quijano E, Pineda R, Marcos S, Yun SH. Brillouin microscopy of collagen crosslinking: noncontact depth-dependent analysis of corneal elastic modulus. Invest Ophthalmol Vis Sci. 2013 Feb 19;54(2):1418-25. doi: 10.1167/iovs.12-11387. PMID 23361513
- [Background] Scarcelli G, Yun SH. In vivo Brillouin optical microscopy of the human eye. Opt Express. 2012 Apr 9;20(8):9197-202. doi: 10.1364/OE.20.009197. PMID 22513631
- [Background] Scarcelli G, Pineda R, Yun SH. Brillouin optical microscopy for corneal biomechanics. Invest Ophthalmol Vis Sci. 2012 Jan 20;53(1):185-90. doi: 10.1167/iovs.11-8281. PMID 22159012
- [Background] Scarcelli G, Yun SH. Confocal Brillouin microscopy for three-dimensional mechanical imaging. Nat Photonics. 2007 Dec 9;2:39-43. doi: 10.1038/nphoton.2007.250. PMID 19812712

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2019-09-23): https://cdn.clinicaltrials.gov/large-docs/22/NCT02118922/Prot_SAP_000.pdf